CLINICAL TRIAL: NCT03209544
Title: A Randomized Controlled Trial on the Effectiveness of an Online Self-help Intervention for Suicidal Ideation
Brief Title: Think Life, an Online Self-help Intervention for Coping With Suicidal Ideation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 2014/1050
Record Dates: First submitted 2017-07-04; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Suicidal Ideation
Keywords: Suicidal ideation; Suicide; Cognitive behavioral therapy; Online intervention
MeSH Terms: conditions — Suicidal Ideation; Suicide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group gains access to Think Life, an online self-help intervention. During 6 weeks they receive a new module on a weekly basis.
  Interventions: Behavioral: Online self-help intervention
- Control group (No Intervention): Waitlist control group. They receive access to Think Life after 12 weeks.

INTERVENTIONS:
Behavioral: Online self-help intervention — The intervention was originally developed by van Spijker, van Straten, and Kerkhof (2010). For this study, it was adapted to the Flemish context and called Think Life. Think Life is mainly based Cognitive Behaviour Therapy (CBT). Additionally, it encompasses elements from Dialectical Behaviour Therapy (DBT), Problem Solving Therapy (PST), and Mindfulness Based Cognitive Therapy (MBCT). It encompasses six modules and every module starts with a psycho-educational section followed by a weekly assignment, core exercises and optional exercises. The participant weekly receives access to a new module. A more detailed description of the intervention is described elsewhere (Kerkhof, van Spijker, & Mokkenstorm, 2013; van Spijker et al., 2010; van Spijker, van Straten, et al., 2014).
  Other Names: Think Life
  Arms: Intervention group

SUMMARY:
The objective of the Think Life study is to test the effect of an online, unguided self-help intervention, i.e. Think Life. The primary hypothesis is that Think Life will reduce suicidal ideation. The secondary hypothesis is that Think Life will lead to improvements in depressive symptoms, hopelessness, rumination, and anxiety. Positive changes are expected after completing Think Life and at follow-up, twelve weeks after baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Have internet access and an e-mail account

Exclusion Criteria:

* No suicidal thoughts (i.e. baseline score on Beck Scale for Suicide Ideation = 0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 724 (Actual)
Dates: Start 2015-04-23 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2016-02-24 (Actual)

PRIMARY OUTCOMES:
Beck Scale for Suicide Ideation | Baseline, and 2, 4, 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in severity of suicidal ideation

SECONDARY OUTCOMES:
Suicidal Ideation Attributes | Baseline, and 2, 4, 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in severity of suicidal ideation
Beck Depression Inventory - second edition | Baseline, and 2, 4, 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in symptoms and severity of depression
Beck Hopelessness Scale | Baseline, and 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in one's negative attitude towards the future
Penn State Worry Questionnaire - Past Week | Baseline, and 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in degree of worrying
Hospital Anxiety and Depression Scale | Baseline, and 6 (post-test) and 12 weeks (follow-up) after baseline
  Changes in anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Kees van Heeringen, MD, PhD, Principal Investigator — Ghent Univeristy - Flemish Centre for Expertise in Suicide Prevention